CLINICAL TRIAL: NCT01394796
Title: Egcg, a dyrk1a Inhibitor as Therapeutic Tool for Reversing Cognitive Deficits in Down Syndrome Individuals.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Rafael de la Torre Fornells, Parc de Salu Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGCG/DYRC1A/DS/IMIM/1
Record Dates: First submitted 2011-07-04; First posted 2011-07-14 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epigallocatechin-3-gallate (EGCG) (Active Comparator): EGCG normally works as a dietary supplement. EGCG administration in Down syndrome patients will result in an improvement of their cognitive performance.A a daily oral dose containing 9 mg/kg (range 6.9-12.7) of EGCG is given during three months.
  Interventions: Dietary Supplement: Epigallocatechin-3-gallate (EGCG)
- Placebo (Placebo Comparator): No active substance is given.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Epigallocatechin-3-gallate (EGCG) — EGCG normally works as a dietary supplement. EGCG administration in Down syndrome patients will result in an improvement of their cognitive performance.A a daily oral dose containing 9 mg/kg (range 6.9-12.7) of EGCG is given during three months.
  Arms: Epigallocatechin-3-gallate (EGCG)
Drug: Placebo — No active treatment is given.
  Arms: Placebo

SUMMARY:
There is a mounting evidence of the modulation properties of the major catechin in green tea, epigallocatechin-3-gallate (EGCG), on dual specificity tyrosine-phosphorylation-regulated kinase 1A (DYRK1A) gene overexpression in the brains of DS mouse models.The aims are to investigate the clinical benefits and safety of EGCG administration in young adults with DS, to establish short-term EGCG effects (three months) on neurocognitive performance, and to determine the persistency or reversibility of EGCG related effects after three months of discontinued use.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed of DS neurological disease, aged between 14-29 years, have given the consent to participate (official custody).

Exclusion Criteria:

* Subjects with neurological disease other than DS, relevant medical disease, co-morbid mental disorder or currently taking any treatment that could interfere with cognitive function or alter any key biomarkers and biochemical parameters analyzed.
* Having suffered from any major illness or undergoing major surgery in the last three months before the study;
* Regular ingestion of medication in the month preceding the study. Exceptions were made for single doses of symptomatic medication administered up to the week preceding the trial.
* Current ingestion of vitamin supplements or catechins or AINE in the two weeks preceding the study.
* History of gastrointestinal, hepatic or renal problems or any other cause that may alter processes of absorption, distribution, metabolism, or excretion of the drug, or that might suggest gastrointestinal irritation to drug.
* Subjects following a vegetarian diet.
* Practice of physical exercise for more than 2 hours per day or energy consume/consumption of more than 3000 kcal per week.

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Memory | Predose baseline and 3 months (end of treatment).
  Memory and learning will be assessed using different neuropsicological tests: Pattern Recognition Memory (PRM), Fuld Object Memory Evaluation (FULD), Paired Associates Learning (PAL).
DYRK1A activity biomarkers | Predose baseline and 3 months (end of treatment).
  Plasma homocysteine (Abbot AxyM),NAD (P)H: quinone oxireductase (NQOI) activity and dyrk1a gene expression in lymphocytes).

SECONDARY OUTCOMES:
Psychomotor speed | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  Motor Screening test (MOT)
Attention | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  Attention will be assessed using the following tests:
  Digit Span: forward recall (from the WMS-III). Spatial Span (SSP): forward recall.
Executive functions | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  Executive functions will be assessed using the following tests:
  Digits Span: backward recall (from the WMS-III). Spatial Span (SSP): backward recall. Word fluency. Intra/Extra dimensional Set Shift (IED)
Visuomotor coordination | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  Visuomotor coordination will be assessed following the these tests:
  Purdue Pegboard Test Visuomotor precision
Functional outcome in daily living and adaptative behaviour | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  Functional outcome in daily living and adaptative behaviour Inventory for Client and Agency Planning (ICAP).
Quality of life | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  Kidscreen-27
Qualitative data on treatment effects | Predose baseline: at 1 month, 3 months (end of treatment) plus 6 months.
  With a brief semi-structured self-made interview